CLINICAL TRIAL: NCT07076654
Title: Effectiveness of Preoperative Oral Caffeine in Preventing Spinal-Induced Hypotension During Cesarean Delivery: A Double Blind Randomized Controlled Trial
Brief Title: Oral Caffeine and Spinal-Induced Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Lecturer of anesthesia and critical care, Cairo University
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Caffeine and hypotension
Record Dates: First submitted 2025-07-01; First posted 2025-07-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-07

CONDITIONS: Spinal Hypotension; Caffeine
Keywords: Spinal hypotension; Caffeine; Cesarean delivery
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Active Comparator): Patients will receive oral caffeine 200 mg before spinal anesthesia
  Interventions: Drug: Caffeine (200 mg)
- Control group (Placebo Comparator): Will receive placebo before spinal anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine (200 mg) — Oral caffeine will be given as 200 mg before spinal anesthesia
  Arms: Caffeine
Drug: Placebo — Patient at this arm will receive placebo
  Arms: Control group

SUMMARY:
Hypotension after spinal anesthesia is critical. Thus several interventions have been proposed to mitigate such effect.

DETAILED DESCRIPTION:
Hypotension is a critical issue related to spinal anesthesia during cesarean delivery. Researchers of this study aimed to evaluate the impact of preoperative oral caffeine on the incidence of spinal hypotension during cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* full term pregnant
* undergoing elective cesarean delivery

Exclusion Criteria:

* patient refusal
* baseline systolic pressure < 100 mmHg
* contraindication to spinal anesthesia
* allergy to caffeine

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-07-12 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Incidence of spinal hypotension | After spinal anesthesia till delivery
  Decrease systolic blood pressure < 20% of baseline value

SECONDARY OUTCOMES:
Time to first hypotensive episode | after induction of spinal anesthesia
  time to incidence of hypotension
Incidence of severe hypotension | After onset of spinal anesthesia
  reduced systolic pressure < 60% of baseline value
APGAR score | at 5 minutes after delivery
  APGAR score calculation at 5 minutes
Umbilical artery pH | At 5 minutes after delivery
  Umbilical artery blood gases

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) will not be shared due to concerns regarding participant privacy and confidentiality. Although data may be de-identified, there remains a risk of re-identification, especially in studies involving small sample sizes or sensitive health information.

REFERENCES:
- [Result] Grosso G, Godos J, Galvano F, Giovannucci EL. Coffee, Caffeine, and Health Outcomes: An Umbrella Review. Annu Rev Nutr. 2017 Aug 21;37:131-156. doi: 10.1146/annurev-nutr-071816-064941. PMID 28826374
- [Result] Antar SS, Metaweh A, Neamatallah H, Abdelfattah M, Abdelbaser I, Awad KA. Preoperative oral caffeine as prophylaxis against post-spinal hypotension in patients undergoing orthopedic lower limb surgery: A randomized, placebo-controlled, double-blinded study. Anaesth Crit Care Pain Med. 2025 Aug;44(4):101537. doi: 10.1016/j.accpm.2025.101537. Epub 2025 May 1. PMID 40318850
- [Result] Helmy MA, Helmy KA, Kaddah RA, Shamma MA, Ali MA, Milad LM. Femoral artery Doppler as a novel predictor of spinal hypotension in elective cesarean delivery cases: a prospective observational study. Int J Obstet Anesth. 2025 Aug;63:104706. doi: 10.1016/j.ijoa.2025.104706. Epub 2025 Jun 18. PMID 40550198
- [Result] Adolf Helmy M, Mansour M, Magdy Milad L, Mohammed Aboelregal E, Magdy Youssef M. Change in femoral artery pulsatility index as a novel predictor of post-spinal anesthesia hypotension in adult patients undergoing infra-umbilical surgeries: A prospective observational study. Anaesth Crit Care Pain Med. 2025 Apr;44(2):101482. doi: 10.1016/j.accpm.2025.101482. Epub 2025 Jan 21. No abstract available. PMID 39848332
- [Result] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Derived] Helmy MA, Helmy KA, Zaki RM, Khatab SA, Embaby SA, Kaddah RA, Shamma MA, Milad LM. Caffeine before cesarean delivery: a novel preventive strategy against spinal hypotension, a double blind placebo-controlled trial. J Anesth Analg Crit Care. 2026 Jan 15. doi: 10.1186/s44158-025-00333-z. Online ahead of print. PMID 41535923